CLINICAL TRIAL: NCT06506084
Title: Observational Study on the Use of Ropeginterferon Alfa-2b in Polycythemia Vera (ROPEG-PV)
Status: Active, not recruiting | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: ROPEG-PV
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b — Data will be collected at each visit during the observational study (total duration: 24 months). In accordance with routine clinical practice in this patient population, visits are expected to take place every 6 months.
  Patients who discontinue ropeginterferon alfa-2b treatment at any time will no longer be followed up.
  Other Names: Besremi

SUMMARY:
Polycythaemia vera (PV) is associated with a reduced quality of life, a high rate of vascular events, and an intrinsic risk of disease evolution. The results of several randomised trials for the treatment with new cytoreductive agents are now available, among which a new ropegylated formulation of interferon alfa-2b (ropeginterferon alfa-2b) have been recently approved in Europe and USA [EMA (2019), FDA (2021) and AIFA (2022)]. The use of this drug in clinical practice is an opportunity for a prospective observational study in a rare disease such as PV; the aim is to evaluate its impact in the practical management of these patients.

Therefore, the main objectives of the present study are to determine:

(i) to what extent ropeginterferon alfa-2b can be prescribed and tolerated in patients with PV; (ii) the risk-benefit of ropeginterferon alfa-2b in patients with PV, followed-up in real-world clinical practice.

DETAILED DESCRIPTION:
Classical Philadelphia-negative myeloproliferative neoplasms (Ph-neg MPNs) including polycythemia vera (PV), essential thrombocythemia (ET), and myelofibrosis (MF) are characterized by uncontrolled clonal proliferation of multipotent bone marrow progenitors, sustained by acquired mutations in JAK2, CALR and MPL genes.

Natural history of PV is marked by life threatening outcomes such as thrombosis, bleeding and clonal evolution towards myelofibrosis and acute myeloid leukemia. Treatment-relevant risk stratification is designed to estimate the likelihood of thrombotic complications, which is estimated to occur before or after diagnosis in 20-30% of patients according disease and patient-related risk factors. The cornerstone of treatment in PV includes scheduled phlebotomy, with a hematocrit (Hct) target of <45% and low-dose aspirin in all patients, regardless of risk category. There is currently broad consensus regarding the need for cytoreductive drugs in high-risk patients with PV identified by age >60 years and prior history of thrombosis.

The results of several andomized trials for the treatment of PV are now available, and, in addition to the standard drug hydroxyurea (HU), both a new ropegylated formulation of interferon alfa-2b3 and ruxolitinib4 are now available have been approved in Europe and US and European LeukemiaNet (ELN) investigators have recently provided recommendations for the use of these drugs in clinical practice in low-risk as well as high-risk patients.

After approval by EMA (2019) and FDA (2021), the drug (ROPEGINTERFERON ALFA-2B) was very recently approved and reimbursed by AIFA (2022) in some subgroups of patients with PV. The use of this drug in clinical practice is an opportunity for a prospective observational study in a rare disease such as PV; the aim is to evaluate its impact in the practical management of these patients, according to Determinazione AIFA 20 marzo 2008 about observational clinical studies, and Decreto Ministeriale 17 dicembre 2004 on non-profit studies.

It is not entirely known which is the percentage of patients who, after careful screening as required in good clinical practice, will fail the indications for concomitant clinical or laboratory abnormalities. Furthermore, the proportion of patients who discontinue the drug during follow-up for intolerance or other reasons is currently unknown and data on the benefit-risk ratio are limited.

Moreover, it should be noted that the haematological and clinical responses obtained in clinical trials not always are replicated in the studies of the real-world clinical practice. In fact, daily management of PV patients does not require the same stringent enrollment and follow-up criteria as instead are necessary in clinical trials. Our proposal may also contribute to better implement the results following the recent guidelines, particularly in some subgroups of patients in which AIFA has established the use with reimbursement by Italian National Health System (NHS) (i.e., patients intolerant to HU, women of childbearing age who plan pregnancy and patients with history of skin cancer).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Polycythemia Vera by WHO 2016
* Patient aged ≥ 18 years old
* Patients in need of cytoreductive treatments with ropeginterferon alfa-2b in first or later lines according to the reimbursability criteria defined by the Italian National Health System
* Patients who have signed the written informed consent for study participation.

Exclusion Criteria:

• Any contraindication for ropeginterferon alfa-2b according to the SmPC

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The first time point to assess the primary outcome defined as the achievement of CHR is after 12 months of treatment with ropeginterferon alfa-2b, is reasonable to provide evidence of at least a non-inferiority in terms of CHR with this new drug. In this framework, a sample size is calculated to test 1-sample non-inferiority of a proportion. Setting the expected proportion p of CHR under ropeginterferon alfa-2b equals to the reference value (p0) obtained with ruxolitinib (i.e., p = p0 = 0.24), a sample size of 319 is needed to demonstrate that the proportion of CHR under ropeginterferon alfa-2b is not inferior to that obtained under ruxolitinib, allowing a margin of non-inferiority (delta) of 0.07 and assuming alpha and beta errors of 5% and 10%, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete hematological remission (CHR)* after 1 and 2 years of treatment. | At baseline and during the follow up at 6/12/18/24 months per patient.
  *HCT lower than 45% without phlebotomies in the past 3 months; platelet count ≤ 400x109/L, WBC count <10 x109/L

SECONDARY OUTCOMES:
Screening failure | At baseline and during the follow up at 6/12/18/24 months per patient.
  Percentage of patients who, after careful screening as required in good clinical practice, will fail the indications for concomitant clinical or laboratory abnormalities.
Complete hematological (CHR) and clinical remission (CR) after 1 and 2 years of treatment stratified by different eligibility categories for treatment indication. | At baseline and during the follow up at 6/12/18/24 months per patient.
  Secondary Outcomes for efficacy
Dose-response effect on CHR and CR | At baseline and during the follow up at 6/12/18/24 months per patient.
  Secondary Outcomes for efficacy
Frequency of phlebotomies | At baseline and during the follow up at 6/12/18/24 months per patient.
  Secondary Outcomes for efficacy
Change in spleen size | At baseline and during the follow up at 6/12/18/24 months per patient.
  Change in spleen size (from baseline) evaluated by palpation.
Incidence of any of the following: o arterial and venous thrombotic events; o hemorrhagic events; o disease related symptoms; o disease evolutions into myelofibrosis and acute leukemia; o secondary malignancies. | At baseline and during the follow up at 6/12/18/24 months per patient.
  Secondary Outcomes for efficacy
Incidence, causality and intensity of any adverse event occurring during study period (as defined by MedDRA code and graded according to Common Terminology Criteria for Adverse Events (CTCAE last version)). | At baseline and during the follow up at 6/12/18/24 months per patient.
  Secondary Outcomes for safety

CONTACTS AND LOCATIONS:
Overall Officials: TIZIANO BARBUI, MD, Study Director — FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS
Locations (37):
- Italy (32):
  - UOC Ematologia, ASST Papa Giovanni XXIII, Bergamo, Lombardy
  - Divisione Ematologia ASST, Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Divisione Ematologia, Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - U.O. Ematologia, Ospedale di Circolo e Fondazione Macchi Varese, Varese, Lombardy
  - Clinica Medica I Azienda Ospedaliera di Padova, Padua, Veneto
  - Divisione Ematologia, Ospedale Borgo Roma, Verona, Veneto
  - Divisione Ematologia, Ospedale San Bortolo, Vicenza, Veneto
  - A.S.O. SS. Antonio e Biagio e C.Arrigo di Alessandria, Alessandria
  - Azienda Ospedaliera Universitaria Consorziale - Policlinico, U.O. Ematologia con Trapianto, Bari
  - Policlinico S. Orsola - Malpighi, Unità di Ematologia, Bologna
  - ASST-Spedali Civili, Brescia
  - Ospedale Businco, S.C. Ematologia e CTMO, Cagliari
  - Azienda Ospedaliero - Universitaria "Policlinico Vittorio Emanuele" - PO Gaspare Rodolico, Dipartimento di Ematologia con Trapianto di midollo Osseo, Catania
  - Azienda Ospedaliera S. Croce e Carle di Cuneo- Divisione di Ematologia,, Cuneo
  - Arcispedale Sant'Anna Azienda Ospedaliero - Universitaria di Ferrara, Unità Operativa di Ematologia, Ferrara
  - Azienda Ospedaliera Universitaria Careggi, Divisione di Ematologia, Florence
  - Azienda Ospedaliera Universitaria Policlinico "G. Martino", UOC Ematologia, Messina
  - Ospedale dell'Angelo, Dipartimento di Ematologia, Mestre
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Ematologia, Milan
  - Ospedale San Raffaele, Unità Operativa di Ematologia e Trapianto Midollo Osseo, Milan
  - ASST MONZA Ospedale San Gerardo Clinica Ematologica, Monza
  - Azienda Ospedaliera Universitaria Federico II di Napoli Divisione di Ematologia e Trapianti del Midollo, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara SCDU Ematologia, Novara
  - Azienda Ospedaliera Universitaria Policlinico "P. Giaccone", Divisione di Ematologia, Palermo
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda Ospedaliera San Eugenio - UOC Ematologia, Roma
  - Fondazione Policlinico Universitario A. Gemelli - Università Cattolica del Sacro Cuore, UCSC Ematologia, Roma
  - Policlinico Umberto I, Dipartimento Ematologia, Oncologia e Dermatologia, Roma
  - Ospedale Casa Sollievo della Sofferenza Istituto di Ricovero e Cura a Carattere Scientifico, U.O. Ematologia, San Giovanni Rotondo
  - A.O.U. Città della Salute e della Scienza di Torino - Ospedale Molinette- S.C. Ematologia U, Torino
  - Ospedale Maggiore, SC Ematologia, Trieste
  - Azienda Sanitaria Universitaria Integrata, Presidio Ospedaliero "Santa Maria della Misericordia", Clinica Ematologica, Udine
- Poland (5):
  - University Medical Center, Department of Hematology and Transplantation, Gdansk
  - Pratia Onkologia, Department of Hematology and Cancer Prevention, Katowice
  - Jagiellonian University Hospital, Department of Haematology, Krakow
  - Copernicus Hospital, Lodz
  - Medical University, Clinical Department of Haematology, Blood Neoplasms and Bone Marrow Transplantation, Wroclaw